CLINICAL TRIAL: NCT03586739
Title: Evaluation of Covered Stents Versus Bare Metal Stents for Endovascular Treatment of Chronic Atherosclerotic Mesenteric Arterial Disease:a Randomised Study.
Brief Title: Evaluation of Covered Stents Versus Bare Metal Stents for Endovascular Treatment of Chronic Ischemia Mesenteric Disease.
Acronym: ESTIMEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0040; 2018-A01833-52 (Other: ID-RCB)
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Mesenteric Ischemia; Stent Stenosis
Keywords: Mesenteric Ischemia Chronic; Atherosclerosis; Restenosis; Primary endovascular treatment; Covered stents; Bare metal stents
MeSH Terms: conditions — Atherosclerosis | interventions — Tomography, X-Ray Computed; Angiography, Digital Subtraction; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Covered stents" strategy (Experimental)
  Interventions: Procedure: endovascular angioplasty using covered stents; Device: Duplex-scan; Device: computerized tomography scan (CT-scan); Device: digital angiography; Other: Short Form-36 (SF-36) questionnaire
- "Bare metal stents" strategy (Active Comparator)
  Interventions: Procedure: endovascular angioplasty using bare metal stents; Device: Duplex-scan; Device: computerized tomography scan (CT-scan); Device: digital angiography; Other: Short Form-36 (SF-36) questionnaire

INTERVENTIONS:
Procedure: endovascular angioplasty using covered stents — Primary endovascular angioplasty using one or several covered stents
  Arms: "Covered stents" strategy
Procedure: endovascular angioplasty using bare metal stents — Primary endovascular angioplasty using one or several bare metal stents
  Arms: "Bare metal stents" strategy
Device: Duplex-scan — a Duplex-scan will be performed during patient follow up.
Device: computerized tomography scan (CT-scan) — a CT-scan will be performed in the event of symptoms of recurrence or restenosis as confirmatory exam according to clinical practice during patient follow up.
  The CT-scan will be mandatory at 12 and 24 months if it has not been planned in the current practice follow-up.
Device: digital angiography — In case CT-scan cannot be performed (e.g. occurrence of a non-preexisting contra-indication), a digital angiography will be authorised instead to confirm restenosis during patient follow-up.
Other: Short Form-36 (SF-36) questionnaire — The patient will complete a quality-of-life questionnaire (SF-36 form) during their follow up.

SUMMARY:
Chronic Mesenteric Ischemia (CMI) is defined by one or more arterial digestive lesions, responsible for severe mesenteric symptoms. The clinical presentation of CMI is characterized by postprandial abdominal pain and weight loss, leading to severe malnutrition. It is a frequent pathology which affects preferentially the elderly patients of female sex (70%) with cardio-vascular comorbidities. Risk factors include smoking, hypertension, and dyslipidemia.

Despite medical and diagnostic advances, the morbidity and mortality of CMI remain very high (>70%). Optimal management of CMI is based on early diagnosis. Symptomatic patients with CMI should be treated without much delay to relief symptoms (present in 43% patients) and prevent acute mesenteric ischemia.

The three visceral arteries affected by atherosclerotic disease are coeliac trunc, inferior mesenteric artery and Superior Mesenteric Artery (SMA). The SMA is treated the most frequently, because it is the main relevant artery associated with CMI.

Endovascular treatment (angioplasty and stenting) is considered as the first-line treatment for CMI when feasible. It is indicated especially in the case of high grade stenosis or occlusion of the Superior Mesenteric Artery. Two types of stents can be used for this procedure: bare metal stents (BMS) or covered stents (CS).

Even if BMS are standard care there is no consensus on the type of stent to use.

There are very few reported series with large numbers of patients comparing BMS and CS in this indication. However, to our knowledge, no results from a randomized study addressing this issue have ever been published. These are only retrospective with a low level of evidence (IIb). The largest series compared 147 patients with primary intervention for CMI treatment using BMS versus 42 using CS. Treatment with CS showed better results in terms of symptom recurrence (10% vs 32%, p <0.002), restenosis (12% vs 42%, p <0.0002) and re-interventions (10% vs 42%), after at least 1 year of follow-up. Indeed, endovascular treatment using BMS was associated with high incidence of symptoms recurrence despite the satisfying patency rates in both occluded and stenotic vessels.

There are no international guidelines to recommend the use of one or another sort of stent.

The necessity of a randomised study addressing the issue of bare metal versus covered stents deployment seems to be important.

The investigators propose to demonstrate that covered stents presents a better efficacy than bare metal stents, with a multicenter randomized study involving 24 vascular surgical departments of French University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Diagnosis of chronic atherosclerotic mesenteric ischemia or atherosclerosis threatening disorders of digestive perfusion, with stenosis or occlusion of the superior mesenteric artery;
* For whom a primary endovascular intervention by percutaneous transluminal angioplasty using stents has been scheduled (anatomical evaluation, arterial evaluation consistent with endovascular treatment);
* For an ostial or post-ostial stenotic arterial lesion to be treated by only one type of stent authorized in the study according to randomization;
* Having signed an informed consent for participation in the study.

Exclusion Criteria:

* Acute mesenteric ischemia;
* Previous revascularisation intervention for chronic mesenteric ischemia;
* For some stenotic arterial lesion to be treated more than one type of stent;
* Chronic renal failure (glomerular filtration rate less than 20 mL per minute);
* Low probability of cooperation of the participant (judged by the investigator);
* Medical or surgical history judged by the investigator to be not compatible with this study;
* Adult ward or court (under guardianship or trusteeship);
* Pregnant or lactating woman;
* Person under judicial protection;
* Subject participating in another study having an exclusion period still active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Freedom from restenosis, | 24 months after the primary endovascular treatment
  Freedom from restenosis will be defined as ≥50% luminal reduction and/or thrombosis, confirmed by CT-scan.
  The crude percentage of restenosis and/or thrombosis at 24 months will be computed for each group. The survival curves for freedom from restenosis and/or thrombosis will be plotted according to the Kaplan-Meier method and overall survival rates will be estimated.

SECONDARY OUTCOMES:
Occurrence of endovascular procedure complications | up to discharge from hospital
Number of patients with maintained primary, primary assisted and secondary patencies | 24 months after the primary endovascular treatment
Number of patients with maintained primary, primary assisted and secondary patencies | 6 months after the primary endovascular treatment
Number of patients with maintained primary, primary assisted and secondary patencies | 12 months after the primary endovascular treatment
Number of patients with maintained primary, primary assisted and secondary patencies | 18 months after the primary endovascular treatment
Target lesion revascularisation (TLR) | 24 months after the primary endovascular treatment
  Repeat revascularisation for a lesion anywhere within the primary stent or the 5-mm borders proximal or distal to the stent
Freedom of symptoms recurrence | 24 months after the primary endovascular treatment
  Clinical recurrence, defined as the symptomatic recurrence of chronic, subacute or acute mesenteric ischemia
Freedom of reintervention (endovascular or surgical) | 24 months after the primary endovascular treatment
Occurrence of major morbidity | 24 months after the primary endovascular treatment
  Occurrence of major morbidity and description of the events
Quality of life score | 24 months after the primary endovascular treatment
  quality of life will be compared between the two groups and assessed using the SF-36 questionnaire
Quality of life score | at inclusion
  quality of life will be compared between the two groups and assessed using the SF-36 questionnaire
Quality of life score | 6 months after the primary endovascular treatment
  quality of life will be compared between the two groups and assessed using the SF-36 questionnaire
Quality of life score | 12 months after the primary endovascular treatment
  quality of life will be compared between the two groups and assessed using the SF-36 questionnaire
Freedom from restenosis | 12 months after the primary endovascular treatment
  The freedom from restenosis will be defined as ≥50% luminal reduction and/or thrombosis, confirmed by CT-scan.
  The crude percentage of restenosis and/or thrombosis at 12 months will be computed for each group. The survival curves for freedom from restenosis and/or thrombosis will be plotted according to the Kaplan-Meier method and overall survival rates will be estimated.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Département de Chirurgie Vasculaire, CHU d'Angers, Angers
  - Département de Chirurgie Vasculaire? CHU J. Minjoz Besançon, Besançon
  - Département de Chirurgie Vasculaire, APHP Hôpital Ambroise Paré, Boulogne-Billancourt
  - Service de Chirurgie Vasculaire, CHU de Brest, Hôpital de La Cavale Blanche, Brest
  - Département de Chirurgie Vasculaire, CHU Clermont-Ferrand - Hôpital G. Montpied, Clermont-Ferrand
  - Département de Chirurgie Cardio-Vasculaire, CHU Le Bocage Dijon Bourgogne, Dijon
  - Département de Chirurgie Vasculaire, CHRU Hôpital Cardiologique de Lille, Lille
  - Département de Chirurgie Vasculaire, Centre Hospitalier Saint Philibert, Lomme, Lomme
  - Département de Chirurgie Vasculaire, CHU Marseille - Hôpital la Timone, Marseille
  - Département de Chirurgie Vasculaire, CHU Nice - Hôpital Pasteur, Nice
  - Département de Chirurgie Vasculaire, APHP Hôpital de la Pitié-Salpêtrière, Paris
  - APHP Hôpital Bichat - Claude Bernard, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - Département de Chirurgie Vasculaire, CHU Poitiers - Hôpital Jean Bernard, Poitiers
  - Département de Chirurgie Vasculaire, CHU Pontchailloux Rennes, Rennes
  - Département de Chirurgie Vasculaire, CHU de Rouen, Rouen
  - Département de Chirurgie Vasculaire, CHU Amiens Picardie - Site Sud, Salouël
  - Service de Chirurgie Vasculaire, CHU de Strasbourg, Nouvel Hôpital Civil, Strasbourg
  - Département de Chirurgie Vasculaire, CHU Toulouse - Hôpital Rangueil, Toulouse
  - Département de Chirurgie Vasculaire? CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy